CLINICAL TRIAL: NCT01751997
Title: The Comparison of Transplantation From Family-mismatched/Haploidentical Donors With Matched Unrelated Donors in Adult Patients With Acute Myeloid Leukemia
Brief Title: Family-mismatched/Haploidentical Donors Versus Matched Unrelated Donors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Byung-Sik Cho (Other)
Responsible Party: Sponsor-Investigator, Byung-Sik Cho, Assistant Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBMTC-AML-1
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transplants from 8/8-matched unrelated (Active Comparator): Participants will receive transplants from 8/8-matched unrelated donors using myeloablative or reduced-intensity conditioning according to age or comorbidity.
  Interventions: Drug: Transplants from 8/8-matched Unrelated donors
- Transplants from family-mismatched/haploidentical donors (Experimental): Participants will receive FMT using a reduced intensity conditioning regimens.
  Interventions: Drug: Transplants from family-mismatched/haploidentical donors

INTERVENTIONS:
Drug: Transplants from 8/8-matched Unrelated donors — * Myeloablative conditioning
    1. Total body irradiation; 165 cGy, every 12 hours, 8 doses, days -7 to -4 (total 1320 cGy)
    2. Cyclophosphamide; 60 mg/kg/day, IV for 30 minutes, days -3 to -2 (total 120 mg/kg)
    3. Antithymocyte globulin (ATG); 1.25 mg/kg/day, IV for 6 hours, days -3 to -2, (total 2.5 mg/kg)
  * Reduced-intensity conditioning; older patients (age > 55 years) and/or patients with comorbidities
    1. Fludarabine; 30 mg/m^2/day, IV for 1 hour, days -8 to -4 (total 150 mg/m^2)
    2. Busulfex; 3.2 mg/kg/day, IV for 3 hours, days -3 to -2 (total 6.4 mg/kg)
    3. Total body irradiation; 200 cGy, every 12 hours 2 doses, days -1 (total 400 cGy)
    4. ATG; 1.25 mg/kg/day, IV for 6 hours, days -3 to -2, (total 2.5 mg/kg)
  * GVHD prophylaxis
    1. Tacrolimus; 0.03 mg/kg/day, IV for 24 hours from day -1 (0.12 mg/kg/day, PO, if tolerable)
    2. Methotrexate; 5 mg/m^2/day, IV push, days +1, +3, +6, +11
  Arms: Transplants from 8/8-matched unrelated
Drug: Transplants from family-mismatched/haploidentical donors — * Reduced-intensity conditioning
    1. Total body irradiation; 200 cGy, every 12 hours, 4 doses, days -9 to -8 (total 800 cGy)
    2. Fludarabine; 30 mg/m^2/day, IV for 1 hour, days -7 to -3 (total 150 mg/m^2)
    3. Busulfex; 3.2 mg/kg/day, IV for 3 hours, days -6 to -5 (total 6.4 mg/kg)
    4. ATG; 1.25 mg/kg/day, IV for 6 hours, days -4 to -1 (total 5.0 mg/kg)
  * GVHD prophylaxis
    1. Tacrolimus; 0.03 mg/kg/day, IV for 24 hours from day -1 (0.12 mg/kg/day, PO, if tolerable)
    2. Methotrexate; 5 mg/m^2/day, IV push, days +1, +3, +6, +11
  Arms: Transplants from family-mismatched/haploidentical donors

SUMMARY:
This study will compare the clinical outcomes of transplants from family-mismatched/haploidentical donors (FMT) with transplants from 8/8-matched unrelated donor (MUT), which is a current gold standard donors when lacking of HLA-matched-siblings

1. Primary objectives: Overall survival of FMT may be similar to that of MUT
2. Secondary objectives:

   i. Comparison of disease-free survival, relapse, non-relapse mortality, immune reconstitution cytomegalovirus infection, and acute or chronic graft-versus-host disease between FMT and MUT.

   ii. Investigation of possible biomarkers related with above events after transplantation

DETAILED DESCRIPTION:
For patients lacking an HLA-identical sibling, 8/8-matched unrelated donors are currently the "gold standard" for a donor, since outcomes after HLA-identical sibling have been compared to 8/8-matched unrelated donors. Currently, there are three alternative graft sources, including mismatched unrelated donors, familial mismatch/haploidentical donors, and umbilical cord bloods. Compared with other sources, transplants from familial mismatch/haploidentical donors (FMT) have the benefit of an immediate availability of a donor, particularly for those patients who urgently need transplantation. Initial reports had characterized FMT to a poor engraftment and a high incidence of graft-versus-host disease. However, outcomes of FMT have significantly improved over the past decade in the optimization of conditioning regimen and graft selection to allow a stable engraftment across major HLA barriers, with promising leukemia-free survival in adults with acute leukemia. Despite the encouraging results and potential benefit of FMT, there have been few studies comparing clinical outcomes of FMT with other donor types, particularly in acute myeloid leukemia (AML) as a single disease. Since August 2008, we have been continuously performing FMT using unmanipulated donor cells and a less aggressive conditioning regimen in high-risk AML lacking an HLA-identical sibling, 8/8 or 7/8-matched unrelated donors. We reported the feasibility of FMT using our novel reduced-intensity regimen without ex vivo T-cell depletion, showing early results similar to outcomes of transplant from 8/8-matched unrelated donors (MUT). This study will test the hypothesis that overall survival at 3 years after FMT is similar to overall survival after MUT.

ELIGIBILITY:
Inclusion Criteria

* Patients with AML aged from 18 to 65 years
* Eastern Cooperative Oncology Group (ECOG) performance < 2
* High risk group for relapse

  1. Complete remission (CR) 1 with unfavorable prognostic factor; presenting white blood cell > 100,000/microliter or prior myelodysplastic syndrome (MDS) or myeloproliferative neoplasm (MPN) or MDS/MPN or cytogenetics & molecular features (intermediate and adverse)
  2. CR2 or CR3 at transplantation
* No HLA-matched sibling and unrelated donor (HLA-A, -B, -C, and -DRB1)
* Acceptable organ function defined as serum creatinine < 2 mg/dl, unless considered due to leukemia and serum bilirubin < 3 mg/dl, unless considered due to leukemia
* Written informed consent form

Exclusion Criteria

* Active uncontrolled infections
* Corrected pulmonary diffusion capacity of <40%
* Cardiac ejection fraction of <35%
* ECOG performance status :2, 3, 4
* Active central nervous system involvement of disease
* Serological evidence of infection with HIV
* Pregnancy or breastfeeding
* Patient who are not suitable for the trial in accordance with principal investigator's decision

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | annually through 3 years
  Overall survival is defined as the time interval between date of enrollment and death from any cause or for surviving patients, to last follow-up

SECONDARY OUTCOMES:
Neutrophil recovery | 56 days
  defined as achieving an absolute neutrophil count greater than or equal to 500/mm^3 for three consecutive measurements on three difference days. The first of the 3 days will be designated the day of neutrophil recovery.
Primary Graft failure | 56 days
  defined as failure to achieve a neutrophil count greater than 500/mm^3 for 3 consecutive days at any time after transplantation.
Secondary Graft failure | 100 days
  defined as the development of an absolute neutrophil count less than 500/mm^3 after achievement of initial engraftment in the absence of recurrent disease.
Platelet recovery | 100 days and 180 days
  defined as the first day of a sustained platelet count greater than 20,000/mm^3 without platelet transfusions in preceding 7 days. The first day of the sustained platelet count will be designated the day of platelet engraftment.
Donor cell engraftment | 56 days
  Donor cell engraftment is defined as donor chimerism greater than or equal 5% on Day 56 after transplantation. Chimerism may be evaluated in whole blood or blood cell fractions, including cluster of differentiation (CD) 3 and CD33 or CD15 fractions. The actual measurement dates may be within +/- 7 days of the above recommended time points.
Acute graft-versus-host disease (aGVHD) | every 3 months through 3 years
  The cumulative incidence of aGVHD (grade II-IV and III-IV) will be determined. The time to onset of aGVHD will be recorded, as well as the maximum grade achieved.
Chronic graft-versus-host disease (cGVHD) | every 3 months through 3 years
  The cumulative incidence of cGVHD will be determined. Data will be collected directly from providers and chart review according to the recommendations of the NIH Consensus Conference. The NIH global severity scores of mild, moderate, and severe cGVHD will be assessed.
Disease free survival | annually through year 3
  defined as the time interval from date of enrollment and time to relapse/progression, to death or to last follow-up
Non-relapse mortality | annually through year 3
  The cumulative incidence of non-relapse mortality will be estimated at Days 100, 180, and at 1 and 2 years after transplantation. An event for this endpoint is death without evidence of disease progression or recurrence
Infection | annually through year 3
  All grade 2 and 3 infections will be reported. Grade 1 cytomegalovirus infections through Day 56 will also be reported.
WT1 MRD assessment | before and 1 month after transplantation, then every 3 months through 3 years
  WT1 MRD assessment
BAALC MRD assessment | before and 1 month after transplantation, then every 3 months through 3 years
  BAALC MRD assessment
NGS-based MRD assessment | before and 1 month after transplantation, then every 3 months through 3 year
  NGS-based MRD assessment
T cells reconstitution | before and 2 weeks and 1 month after transplantation, then every 3 months through 1 year
  T cell subsets
NK cells reconstitution | before and 2 weeks and 1 month after transplantation, then every 3 months through 1 year
  NK cell subsets
B cells reconstitution | before and 2 weeks and 1 month after transplantation, then every 3 months through 1 year
  B cells

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Je Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hematology Hospital
Locations (1):
- Catholic Blood and Marrow Transplantation Center, Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Background] Aversa F. Haploidentical haematopoietic stem cell transplantation for acute leukaemia in adults: experience in Europe and the United States. Bone Marrow Transplant. 2008 Mar;41(5):473-81. doi: 10.1038/sj.bmt.1705966. Epub 2008 Jan 7. PMID 18176612
- [Background] Ruggeri A, Ciceri F, Gluckman E, Labopin M, Rocha V; Eurocord and Acute Leukemia Working Party of the European Blood and Marrow Transplant Group. Alternative donors hematopoietic stem cells transplantation for adults with acute myeloid leukemia: Umbilical cord blood or haploidentical donors? Best Pract Res Clin Haematol. 2010 Jun;23(2):207-16. doi: 10.1016/j.beha.2010.06.002. PMID 20837332
- [Background] Yakoub-Agha I, Mesnil F, Kuentz M, Boiron JM, Ifrah N, Milpied N, Chehata S, Esperou H, Vernant JP, Michallet M, Buzyn A, Gratecos N, Cahn JY, Bourhis JH, Chir Z, Raffoux C, Socie G, Golmard JL, Jouet JP; French Society of Bone Marrow Transplantation and Cell Therapy. Allogeneic marrow stem-cell transplantation from human leukocyte antigen-identical siblings versus human leukocyte antigen-allelic-matched unrelated donors (10/10) in patients with standard-risk hematologic malignancy: a prospective study from the French Society of Bone Marrow Transplantation and Cell Therapy. J Clin Oncol. 2006 Dec 20;24(36):5695-702. doi: 10.1200/JCO.2006.08.0952. Epub 2006 Nov 20. PMID 17116940
- [Background] Beatty PG, Clift RA, Mickelson EM, Nisperos BB, Flournoy N, Martin PJ, Sanders JE, Stewart P, Buckner CD, Storb R, et al. Marrow transplantation from related donors other than HLA-identical siblings. N Engl J Med. 1985 Sep 26;313(13):765-71. doi: 10.1056/NEJM198509263131301. PMID 3897863
- [Background] Anasetti C, Hansen JA. Effect of HLA incompatibility in marrow transplantation from unrelated and HLA-mismatched related donors. Transfus Sci. 1994 Sep;15(3):221-30. doi: 10.1016/0955-3886(94)90134-1. PMID 10155543
- [Background] Henslee-Downey PJ, Abhyankar SH, Parrish RS, Pati AR, Godder KT, Neglia WJ, Goon-Johnson KS, Geier SS, Lee CG, Gee AP. Use of partially mismatched related donors extends access to allogeneic marrow transplant. Blood. 1997 May 15;89(10):3864-72. PMID 9160695
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Ruggeri L, Mancusi A, Capanni M, Urbani E, Carotti A, Aloisi T, Stern M, Pende D, Perruccio K, Burchielli E, Topini F, Bianchi E, Aversa F, Martelli MF, Velardi A. Donor natural killer cell allorecognition of missing self in haploidentical hematopoietic transplantation for acute myeloid leukemia: challenging its predictive value. Blood. 2007 Jul 1;110(1):433-40. doi: 10.1182/blood-2006-07-038687. Epub 2007 Mar 19. PMID 17371948
- [Background] Ciceri F, Labopin M, Aversa F, Rowe JM, Bunjes D, Lewalle P, Nagler A, Di Bartolomeo P, Lacerda JF, Lupo Stanghellini MT, Polge E, Frassoni F, Martelli MF, Rocha V; Acute Leukemia Working Party (ALWP) of European Blood and Marrow Transplant (EBMT) Group. A survey of fully haploidentical hematopoietic stem cell transplantation in adults with high-risk acute leukemia: a risk factor analysis of outcomes for patients in remission at transplantation. Blood. 2008 Nov 1;112(9):3574-81. doi: 10.1182/blood-2008-02-140095. Epub 2008 Jul 7. PMID 18606875
- [Background] Huang XJ, Liu DH, Liu KY, Xu LP, Chen H, Han W, Chen YH, Zhang XH, Lu DP. Treatment of acute leukemia with unmanipulated HLA-mismatched/haploidentical blood and bone marrow transplantation. Biol Blood Marrow Transplant. 2009 Feb;15(2):257-65. doi: 10.1016/j.bbmt.2008.11.025. PMID 19167686
- [Background] Cho BS, Yoon JH, Shin SH, Yahng SA, Lee SE, Eom KS, Kim YJ, Lee S, Min CK, Cho SG, Kim DW, Lee JW, Min WS, Park CW, Kim HJ. Comparison of allogeneic stem cell transplantation from familial-mismatched/haploidentical donors and from unrelated donors in adults with high-risk acute myelogenous leukemia. Biol Blood Marrow Transplant. 2012 Oct;18(10):1552-63. doi: 10.1016/j.bbmt.2012.04.008. Epub 2012 Apr 16. PMID 22516055
- [Derived] Cho BS, Min GJ, Park S, Park SS, Shin SH, Yahng SA, Jeon YW, Yoon JH, Lee SE, Eom KS, Kim YJ, Lee S, Min CK, Cho SG, Kim DW, Lee JW, Kim M, Kim Y, Kim HJ. Haploidentical vs matched unrelated donor transplantation for acute myeloid leukemia in remission: A prospective comparative study. Am J Hematol. 2021 Jan;96(1):98-109. doi: 10.1002/ajh.25993. Epub 2020 Nov 24. PMID 32905642